CLINICAL TRIAL: NCT02822937
Title: A Study to Assess the Sensitivity of Project: EVO Monitor Cognitive Function Measurements to Methylphenidate and Triazolam in Adults 40-55 Years Old
Brief Title: Sensitivity of Project: EVO Monitor Cognitive Measurements to Pharmacological Agents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akili Interactive Labs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: Akili-027
Record Dates: First submitted 2016-06-02; First posted 2016-07-06 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Healthy
MeSH Terms: interventions — Methylphenidate; Triazolam; Sugars

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo, Methylphenidate, Triazolam (Experimental): The participants will receive placebo on the first day, 40mg Methylphenidate on the second day, and 0.375mg Triazolam on the third day. All drug administration and cognitive measurement will take place in the clinic under medical staff supervision. During each study day in the clinic, the participants will use Project: EVO Monitor and do a short digit symbol substitution task (DSST) 8 times over the day.
  Interventions: Drug: Methylphenidate; Drug: Triazolam; Other: Project: EVO; Drug: Placebo
- Placebo, Triazolam, Methylphenidate (Experimental): The participants will receive placebo on the first day, 0.375mg Triazolam on the second day, and 40mg Methylphenidate on the third day. All drug administration and cognitive measurement will take place in the clinic under medical staff supervision. During each study day in the clinic, the participants will use Project: EVO Monitor and do a short digit symbol substitution task (DSST) 8 times over the day.
  Interventions: Drug: Methylphenidate; Drug: Triazolam; Other: Project: EVO; Drug: Placebo
- Methylphenidate, Placebo, Triazolam (Experimental): The participants will receive 40mg Methylphenidate on the first day, placebo on the second day, and 0.375mg Triazolam on the third day. All drug administration and cognitive measurement will take place in the clinic under medical staff supervision. During each study day in the clinic, the participants will use Project: EVO Monitor and do a short digit symbol substitution task (DSST) 8 times over the day.
  Interventions: Drug: Methylphenidate; Drug: Triazolam; Other: Project: EVO; Drug: Placebo
- Methylphenidate, Triazolam, Placebo (Experimental): The participants will receive 40mg Methylphenidate on the first day, 0.375mg Triazolam on the second day, and placebo on the third day. All drug administration and cognitive measurement will take place in the clinic under medical staff supervision. During each study day in the clinic, the participants will use Project: EVO Monitor and do a short digit symbol substitution task (DSST) 8 times over the day.
  Interventions: Drug: Methylphenidate; Drug: Triazolam; Other: Project: EVO; Drug: Placebo
- Triazolam, Placebo, Methylphenidate (Experimental): The participants will receive 0.375mg Triazolam on the first day, placebo on the second day, and 40mg Methylphenidate on the third day. All drug administration and cognitive measurement will take place in the clinic under medical staff supervision. During each study day in the clinic, the participants will use Project: EVO Monitor and do a short digit symbol substitution task (DSST) 8 times over the day.
  Interventions: Drug: Methylphenidate; Drug: Triazolam; Other: Project: EVO; Drug: Placebo
- Triazolam, Methylphenidate, Placebo (Experimental): The participants will receive 0.375mg Triazolam on the first day, 40mg Methylphenidate on the second day, and placebo on the third day. All drug administration and cognitive measurement will take place in the clinic under medical staff supervision. During each study day in the clinic, the participants will use Project: EVO Monitor and do a short digit symbol substitution task (DSST) 8 times over the day.
  Interventions: Drug: Methylphenidate; Drug: Triazolam; Other: Project: EVO; Drug: Placebo

INTERVENTIONS:
Drug: Methylphenidate — Methylphenidate is a central nervous system stimulant. It affects chemicals in the brain and nerves that contribute to hyperactivity and impulse control. Methylphenidate is used to treat attention deficit disorder (ADD), attention deficit hyperactivity disorder (ADHD), and narcolepsy.
  Other Names: Ritalin
Drug: Triazolam — Triazolam is a benzodiazepine similar to Valium. Triazolam affects chemicals in the brain that may become unbalanced and cause sleep problems (insomnia). Triazolam is used to treat insomnia (trouble falling or staying asleep).
  Other Names: Halcion
Other: Project: EVO — Project: EVO Monitor was designed to incorporate a proprietary multi-tasking assessment into a state-of-the-art mobile video game-like platform, which deploys modern videogame graphics, engaging reward loops, and real-time adaptive mechanics to dynamically personalize difficulty in order to assess the user's ability.
  Other Names: Cognitive Monitor
Drug: Placebo — Sugar pill
  Other Names: Sugar Pill

SUMMARY:
This is a study in adults to assess the sensitivity of Project: EVO Monitor cognitive measurements to two short-acting cognitively active pharmacological agents. The participants will receive a placebo, and two pharmacological agents in a randomized order for three in-clinic study days. During each study day in the clinic, the participants will use Project: EVO Monitor and another cognitive task through the day.

DETAILED DESCRIPTION:
This is a study in adults ages 40 to 55 to assess the sensitivity of Project: EVO Monitor cognitive measurements to two short-acting cognitively active pharmacological agents, methylphenidate (MPH) and triazolam (TRZ). The participants will receive a placebo, MPH, and TRZ in a randomized order for three in-clinic study days. All drug administration and cognitive testing will take place in the clinic under medical staff supervision. During each study day in the clinic, the participants will use Project: EVO Monitor and do a short digit symbol substitution task (DSST) 8 times over the day. A minimum of 48 hours will be needed between each study day. The investigators plan to evaluate 18 participants in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-55 at the time of informed consent
2. Ability to follow written and verbal instructions (English).
3. Weight between 140 lbs and 240 lbs.
4. Male and female (Gender-matched).
5. Ability to comply with all the testing and requirements.

Exclusion Criteria:

1. Known adverse reaction to study medications.
2. Known non-response or paradoxical response to study medications.
3. Current, controlled (requiring a restricted medication) or uncontrolled, self-reported psychiatric diagnosis with significant symptoms such as post-traumatic stress disorder, psychosis, bipolar illness, pervasive developmental disorder, severe obsessive compulsive disorder, severe depressive or anxiety disorder, conduct disorder, attention deficit disorder, autism spectrum disorder, or other symptomatic manifestations that in the opinion of the Investigator that may confound study data/assessments.
4. Current self-reported community diagnosis of cognitive ailments such as dementia, Alzheimer's disease, stroke, traumatic brain injury, or other diseases that in the opinion of the Investigator that may confound study data/assessments.
5. Current diagnosis of severe learning disorder, dyslexia, or dyscalculia.
6. Current subjective complaints of inattention or memory loss.
7. Currently undergoing psychotherapy, behavioral therapy, or occupational therapy.
8. Current use of psychotropic medication, prescription or otherwise.
9. Motor condition that prevents game playing, as reported by parent or observed by investigator.
10. Impaired visual acuity, as defined by difficulty reading the informed consent even with corrective lenses.
11. Lifetime history of suspected substance abuse or dependence.
12. Current use (defined as within the last 30 days) of products with nicotine, e.g. cigarettes, chewing tobacco, e-cigarettes, nicotine patch, and nicotine gum.
13. History of seizures (exclusive of febrile seizures), a tic disorder, significant tics, a current diagnosis of Tourette's Disorder.
14. Taken part in a clinical trial within 30 days prior to screening.
15. Diagnosis of or patient-reported color blindness.
16. Regular use of psychoactive drugs that in the opinion of the Investigator may confound study data/assessments.
17. Pregnancy.
18. Currently nursing or breastfeeding.
19. Resting heart rate > 100 beats/min.
20. Systolic blood pressure > 150 mm/Hg.
21. History of cardiac abnormalities.
22. History of glaucoma.
23. Current use of monoamine oxidase inhibitors, HIV protease inhibitors, ranitidine, isoniazid, ketoconazole, itraconazole, nefazodone and other azole-type antifungal agents or any other drugs that are contra-indicated for use with study medications.
24. Any other medical condition that in the opinion of the investigator may confound study data/assessments.
25. Any other medical condition that in the opinion of the investigator prohibits the administration of any study medication.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-07; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Intra-subject sensitivity of Project: EVO cognitive measurements (threshold based) to a cognitive enhancer or a cognitive disruptor at peak drug effects relative to placebo | Measurements taken 120 min post drug with a comparison between 3 clinic visits (each with different drug) over 2 weeks
Intra-subject sensitivity of Project: EVO cognitive measurements (reaction time based) to a cognitive enhancer or a cognitive disruptor at peak drug effects relative to placebo | Measurements taken 120 min post drug with a comparison between 3 clinic visits (each with different drug) over 2 weeks

SECONDARY OUTCOMES:
Intra-subject sensitivity of Project: EVO cognitive measurements (threshold based) to the cognitive enhancer and cognitive disruptor relative to the placebo measurements using the area-under-the-curve (AUC) analysis | Measurements taken predose and 30, 60, 90, 120, 150, 180, and 240 min post drug with a comparison between 3 clinic visits (each with different drug) over 2 weeks
Intra-subject sensitivity of Project: EVO cognitive measurements (reaction time based) to the cognitive enhancer and cognitive disruptor relative to the placebo measurements using the area-under-the-curve (AUC) analysis | Measurements taken predose and 30, 60, 90, 120, 150, 180, and 240 min post drug with a comparison between 3 clinic visits (each with different drug) over 2 weeks
Intra-subject sensitivity to Project: EVO cognitive measurements (threshold based) with the onset and decline of the predicted drug effects over the study day, using a quadratic regression model | Measurements taken predose and 30, 60, 90, 120, 150, 180, and 240 min post drug with a comparison between 3 clinic visits (each with different drug) over 2 weeks
Intra-subject sensitivity to Project: EVO cognitive measurements (reaction time based) with the onset and decline of the predicted drug effects over the study day, using a quadratic regression model | Measurements taken predose and 30, 60, 90, 120, 150, 180, and 240 min post drug with a comparison between 3 clinic visits (each with different drug) over 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ted Riley, Study Director — ProMedica International
Locations (1):
- Clinical Trials of Texas, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No